CLINICAL TRIAL: NCT00873613
Title: Digital Ocular Fundus Photography in the Emergency Department: A New Application for Telemedicine?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Beau Bruce, MD, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: IRB00006900
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Headache; Acute, Focal Neurologic Disease; Severely Elevated Blood Pressure; Acute Visual Loss
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct ophthalmoscopy (No Intervention)
- Non-dilated retinal photography (Experimental)
  Interventions: Procedure: Use of Non-dilated retinal photography

INTERVENTIONS:
Procedure: Use of Non-dilated retinal photography — Kowa Non-Myd alpha-D Non-dilated fundus camera will be used to obtain photographs.
  Arms: Non-dilated retinal photography

SUMMARY:
The purpose of this study is to determine if non-dilated retinal photography in the emergency room improves the diagnosis of papilledema (optic nerve swelling) in patients with neurologic disease compared to direct ophthalmoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Presenting complaint of headache, acute focal neurologic disease, or acute visual changes
* Diastolic blood pressure >= 120
* Age 18 or older

Exclusion Criteria:

* Unable to sit-up, not interested in participation, confused
* Age 17 or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference in detection rate of papilledema by emergency department physicians using non-dilated retinal photography vs. direct ophthalmoscopy. | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Bruce BB, Lamirel C, Wright DW, Ward A, Heilpern KL, Biousse V, Newman NJ. Nonmydriatic ocular fundus photography in the emergency department. N Engl J Med. 2011 Jan 27;364(4):387-9. doi: 10.1056/NEJMc1009733. No abstract available. PMID 21268749
- [Result] Bruce BB, Lamirel C, Biousse V, Ward A, Heilpern KL, Newman NJ, Wright DW. Feasibility of nonmydriatic ocular fundus photography in the emergency department: Phase I of the FOTO-ED study. Acad Emerg Med. 2011 Sep;18(9):928-33. doi: 10.1111/j.1553-2712.2011.01147.x. PMID 21906202
- [Result] Bruce BB, Thulasi P, Fraser CL, Keadey MT, Ward A, Heilpern KL, Wright DW, Newman NJ, Biousse V. Diagnostic accuracy and use of nonmydriatic ocular fundus photography by emergency physicians: phase II of the FOTO-ED study. Ann Emerg Med. 2013 Jul;62(1):28-33.e1. doi: 10.1016/j.annemergmed.2013.01.010. Epub 2013 Feb 21. PMID 23433654